CLINICAL TRIAL: NCT05506904
Title: Liberation From Mechanical Ventilation Using Extubation Advisor Decision Support: The Multicentre (LEADS) Pilot Trial
Brief Title: Liberation From Mechanical Ventilation Using Extubation Advisor Decision Support
Acronym: LEADS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EA-LEADS-001
Record Dates: First submitted 2022-08-02; First posted 2022-08-18 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Airway Extubation

STUDY DESIGN:
Intervention Model Description: Multicentre pragmatic vanguard pilot RCT of the EA tool in invasive ventilated critically ill patients, with and without COVID-19. Individual patients will be randomized (1:1) to intervention (EA tool) or control (standard care).
Who Masked: Outcomes Assessor
Masking Description: Statisticians will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extubation Advisor (Experimental): Wave form data from participants' spontaneous breathing trials (SBT) will be analyzed using Extubation Advisor (EA) to generate an EA report that provides clinical decision support regarding extubation.
  Interventions: Device: Extubation Advisor
- Standard of Care Arm (No Intervention): Participants will undergo SBTs as directed by clinicians. The EA device will not be used.

INTERVENTIONS:
Device: Extubation Advisor — Participants undergoing a Spontaneous Breathing Trial (SBT) to assess readiness for extubation will be connected to a portable monitor displaying ECG, capnography, and other waveforms. This monitor will also be connected to a laptop containing the Extubation Advisor (EA) software. During the SBT, relevant patient information will be entered into the EA application and the EA application will record waveform data. When the SBT is complete, the EA application will analyze the waveform and patient data to generate a score summarizing the risk of extubation failure. A report will be generated and provided to the respiratory therapist and attending physician to help determine whether to proceed with extubation or not. The clinical outcome case report form will be completed at the time of hospital discharge.
  Arms: Extubation Advisor

SUMMARY:
Timely and safe extubation in critically ill patients is vitally important as prolonged mechanical ventilation and failed attempts at extubation are associated with increased morbidity, mortality, costs, intensive care unit (ICU) stays, and a risk for aerosolization of COVID-19 to health care providers. A Spontaneous Breathing Trial (SBT) is the current standard of care to assess a patient's readiness for extubation. However, SBTs are performed in various ways and have poor ability to predict successful extubation on their own. There is an urgent need to improve and standardize extubation decision-making. In a prior multicenter study, the investigators showed that decreased respiratory rate variability during SBTs predicted extubation failure better than other predictive indices.

The Extubation Advisor (EA) tool combines clinician's assessments of extubation readiness with predictive analytics and risk mitigation strategies for individual patients. In a single centre observational study, the investigators demonstrated the ability to deliver EA reports to the bedside and acceptability of this decision-support tool to respiratory therapists (RTs) and physicians (MDs).

The investigators will conduct the Liberation from mechanical ventilation using EA Decision Support (LEADS) Pilot Trial to assess feasibility outcomes. They will include critically ill adults who are invasively ventilated for >48 hours and are ready to undergo an SBT.

Patients in the intervention arm undergo an EA assessment and treating clinicians (RTs, MDs) will receive an EA report for each SBT conducted. The EA report will help to guide extubation decision-making. Patients in the control arm receive standard care. SBTs will be directed by clinicians.

The primary feasibility outcome will reflect the ability to recruit the desired population. The investigators will also assess the usefulness of the tool to MDs and complete an analysis of resource utilization to inform future economic analyses of cost-effectiveness. The investigators aim to recruit 1 to 2 patients/month/center.

The LEADS trial is novel and low-risk. It is the first trial to evaluate use of a bedside decision support tool to assist ICU clinicians with extubation decision-making. The LEADS pilot trial will inform the design of a future, large-scale randomized controlled trial that is expected to enhance the care delivered to critically ill patients, improve extubation outcomes, and inform extubation practice in ICUs.

DETAILED DESCRIPTION:
Background: Timely and safe extubation (i.e. endotracheal tube removal) in critically ill patients is vitally important as prolonged mechanical ventilation and failed attempts at extubation (i.e. re-intubation<48 hrs; 15% incidence) are associated with increased morbidity, mortality, costs, intensive care unit (ICU) stays, and a risk for aerosolization of COVID-19 to health care providers. A Spontaneous Breathing Trial (SBT) is the current standard of care to assess a patient's readiness for extubation. However, SBTs are performed in various ways and have poor ability to predict successful extubation on their own. There is an urgent need to improve and standardize extubation decision-making in the intensive care unit. In a prior multicenter study (n=721), the investigators showed that decreased respiratory rate variability during SBTs predicted extubation failure better than other predictive indices. The Extubation Advisor (EA) tool combines clinician's assessments of extubation readiness with predictive analytics and risk mitigation strategies for individual patients. In a single centre observational study (n=117; 2 ICUs), the investigators demonstrated the ability to deliver EA reports to the bedside and acceptability of this decision-support tool to respiratory therapists (RTs) and physicians (MDs).

Proposed Trial: The investigators will conduct the Liberation from mechanical ventilation using EA Decision Support (LEADS) Pilot Trial to assess feasibility outcomes including recruitment of critically ill patients with and without COVID-19 and protocol adherence.

Patients: The investigators will include critically ill adults who are invasively ventilated for >48 hours and who are ready to undergo an SBT with a view to extubation.

Intervention: Patients in the intervention arm will undergo an EA assessment and treating clinicians (RTs, MDs) will receive an EA report for each SBT conducted. The EA report will help to guide, rather than direct extubation decision-making by MDs.

Control: Patients in the control arm will receive standard care. SBTs will be directed by clinicians, using current best evidence. No EA assessments will be made, and no EA reports will be generated.

Outcomes: The primary feasibility outcome will reflect the ability to recruit the desired population. Secondary feasibility outcomes will assess rates of (i) consent (for eligible patients approached), (ii) randomization, (iii) intervention adherence, (iv) crossovers (EA to standard care and standard care to EA), and (v) completeness of clinical outcomes collected. The investigators will also assess the usefulness of the tool to MDs and complete an analysis of resource utilization to inform future economic analyses of cost-effectiveness. The investigators aim to recruit 1 to 2 patients/month/center on average. The investigators aim to achieve >75% consent rate, >95% randomization rate in consented patients, >80% of EA reports generated and delivered (intervention arm), <10% crossovers (both arms), and >90% of patients with complete clinical outcomes. The investigators will report feasibility outcomes overall and by site.

Impact: The LEADS trial was informed by extensive preparatory work conducted within two parallel programs of research on weaning and extubation. The LEADS trial is novel and low-risk. It is the first trial to evaluate use of a bedside decision support tool to assist ICU clinicians with extubation decision-making. The LEADS pilot trial will inform the design of a future, large-scale randomized controlled trial that is expected to enhance the care delivered to critically ill patients, improve extubation outcomes, and inform extubation practice in ICUs.

ELIGIBILITY:
Inclusion Criteria:

* With or without COVID-19
* In the intensive care unit (ICU)
* Able to provide informed consent (through a surrogate)
* Critically ill adults (age≥18)
* Anticipated to need invasive ventilation for >48 hours prior to an initial SBT
* Ready to undergo an initial SBT within the next 24 hours with a view to extubation as per treating MDs. As per the FAST trial, an SBT will be defined as a focused assessment on low ventilator settings [T-piece, continuous positive airway pressure (CPAP), or PS < 8 cm H2O regardless of positive end-expiratory pressure (PEEP)]

Exclusion Criteria:

* Suffer from known or suspected peripheral severe myopathy or neuropathy, or limb weakness or paralysis or central (e.g., post arrest, large intracranial stroke or bleed) injury or Glasgow Coma Scale (GCS) < 6
* Do not wish to be re-intubated as part of their treatment goals
* Were previously extubated during the same ICU admission
* Have undergone 1 or more SBTs
* Already have a tracheostomy
* Are moribund or expected to die.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of enrolling 1-2 patients per centre per month | Upon study completion, 12 months after study initiation
  Feasibility of patient enrolment will be evaluated by determining if 1-2 patients are enrolled per centre per month.

SECONDARY OUTCOMES:
Evaluate feasibility of consenting greater than 75% of eligible patients | Upon study completion, 12 months after study initiation
  Feasibility of consenting eligible patients will be evaluated by determining if greater than 75% of eligible patients are consented to participate.
Evaluate feasibility of randomizing greater the 95% of consented patients | Upon study completion, 12 months after study initiation
  Feasibility of randomizing consented patients will be evaluated by determining if greater than 95% of consented patients are randomized to either the intervention or standard of care arm.
Evaluate feasibility of generating and delivering greater than 80% of EA reports to the attending physician | Upon study completion, 12 months after study initiation
  Feasibility of EA report generation will be evaluated by determining if greater than 80% of the time, EA reports are generated and delivered to the attending physician.
Evaluate feasibility of crossovers between the intervention and control arms occurring less than 10% of the time | Upon study completion, 12 months after study initiation
  Feasibility of limiting crossovers will be evaluated by determining if crossovers between the intervention and control arms occur less than 10% of the time.
Evaluate feasibility of collecting complete patient outcomes greater than 90% of the time | Upon study completion, 12 months after study initiation
  Feasibility of collecting complete patient outcomes will be evaluated by determining if complete patient outcomes are collected greater than 90% of the time.
Evaluate usefulness of EA reports | Upon study completion, 12 months after study initiation
  Usefulness of EA reports will be evaluated by MDs using a Likert scale (1-6) and be evaluated overall, by centre, by MD experience, and by MD gender. The minimum value of the scale (1) will be "not useful" and the maximum value of the scale (6) will be "very useful", with a higher value indicating a more positive opinion of the EA report.
Evaluate institutional costs required to implement the EA device | Upon study completion, 12 months after study initiation
  The institutional costs required to implement the EA device will be evaluated by collecting institutional costs.
Evaluate the time required by respiratory therapists to implement the EA device | Upon study completion, 12 months after study initiation
  The time required by respiratory therapists to implement the EA device will be evaluated by collecting the amount of time respiratory therapist spend implementing the EA device.
Evaluate the time required by research coordinators to implement the EA device | Upon study completion, 12 months after study initiation
  The time required by research coordinators to implement the EA device will be evaluated by collecting the amount of time research coordinators spend implementing the EA device.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Burns, MD PhD FRCSC, Principal Investigator — Unity Health Toronto - St. Michael's Hospital
Locations (12):
- Canada (12):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Kingston Health Sciences Centre, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Queensway Carleton Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Unity Health Toronto - St. Michael's Hospital, Toronto, Ontario
  - Hotel Dieu de Levis, Lévis, Quebec
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Hopital de l'Enfant Jesus, Québec, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Ste-Foy, Quebec

IPD SHARING:
Plan to Share IPD: Yes
The authors will make the trial data available in a de-identified format upon submission, review and approval of a written request and study outline. This may include all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This information will be available 4 months after pilot trial completion (estimated Oct 2025) and for 5 years thereafter.
Access Criteria: Data will be provided for secondary analyses or data syntheses ( e.g., meta-analyses) accompanied by a study protocol and ethics approval. The authors reserve the write to withhold data related to treatment allocation should the patients in the pilot trial be rolled forward into a larger trial. Drs. Burns and Seeky will review requests for access to deidentified data.

REFERENCES:
- [Derived] Burns KEA, Allan JE, Lee E, Santos-Taylor M, Kay P, Greco P, Every H, Mooney O, Tanios M, Tan E, Herry CL, Scales NB, Gouskos A, Tran A, Iyengar A, Maslove DM, Kutsogiannis J, Charbonney E, Mendelson A, Lellouche F, Lamontagne F, Scales D, Archambault P, Turgeon AF, Seely AJE, Group CCCT. Liberation from mechanical ventilation using Extubation Advisor Decision Support (LEADS): protocol for a multicentre pilot trial. BMJ Open. 2025 Mar 18;15(3):e093853. doi: 10.1136/bmjopen-2024-093853. PMID 40107679